CLINICAL TRIAL: NCT03488706
Title: Assessing Circulating Tumor Cell as a Biomarker for Prostate Cancer Detection in Patients With Gray Zone PSA Level
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CellMaxLife (Industry)
Responsible Party: Sponsor
Other Study IDs: CMx-CTC-PC-001
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gray Zone Group: The gray zone group PSA between 4.00 to 10.99 ng/ml.

SUMMARY:
Prostate cancer screening with PSA is plagued by high rate of unnecessary prostate biopsies, especially in the "gray zone" (4.00ng/ml e 10.99ng/ml). We introduce a new circulating-tumor-cell (CTC) biomarker for detection of prostate cancer in patients in the PSA "gray zone" level, with the clinically verified potential to substantially decrease the number of unnecessary prostate biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are willing to sign the informed consent and agree to comply with the study procedures.
* Age from 20 to 99 years old
* Subjects with a PSA 4.00- 10.99 ng/ml and will receive biopsy within 3 months

Exclusion Criteria:

* Age < 20 years
* Refuse to sign the informed consent form
* Received regional anesthesia and general anesthesia within one month
* Previous cancer history
* Autoimmune diseases
* Chronic inflammatory diseases
* Diagnosed with colorectal polyps or adenomas
* Acute inflammatory or infectious diseases in three months
* Other diseases decided by PI

Ages: 20 Years to 99 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: PSA 4.00- 10.99 ng/ml patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-12-12 (Estimated); Study Completion 2021-06-02 (Estimated)

PRIMARY OUTCOMES:
Circulating tumor cells detection | Prior to prostate biopsy
  Using a circulating-tumor-cell (CTC) test to detect prostate cancer in patients in the PSA "gray zone" level

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Hsu Chang, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan